CLINICAL TRIAL: NCT03954457
Title: Social Ecology and the Prevention of Suicide and Aggression in African American Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePaul University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, LaVome Robinson, Professor of Psychology, DePaul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LR052913PSY; R01HD072293 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Suicide; Aggression
Keywords: Suicide; Aggression; Prevention; Culturally-Adapted; African American Adolescents
MeSH Terms: conditions — Suicide; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-CWS Intervention (Experimental): Participants received A-CWS Intervention.
  Interventions: Behavioral: A-CWS
- Standard Care Control (Active Comparator): Participants received standard care.
  Interventions: Behavioral: Standard Care Control

INTERVENTIONS:
Behavioral: A-CWS — The A-CWS intervention is a 15-session culturally-grounded, cognitive-behavioral group intervention designed to develop and enhance African American youths' skills for coping with stress. The intervention structure allows implementation within traditional school and other community settings. The A-CWS uses standard cognitive-behavioral strategies (e.g., relaxation training, cognitive restructuring) to help African American youth identify and cope with individual and contextual stressors, using culturally consistent coping strategies. The intervention emphasizes the identification and management of stressors associated with suicide risk (e.g., racism-related stress, community violence exposure) and the unique experiences of low-resourced, urban African American adolescents (e.g., community violence exposure). The structured, manualized A-CWS curriculum is designed to be sustainable and user-friendly, to ensure that the A-CWS is delivered effectively and with a high degree of fidelity.
  Arms: A-CWS Intervention
Behavioral: Standard Care Control — The standard care control condition consisted of standard case management services delivered by the SBHC. Participants randomly assigned to the standard care control condition were referred to the SBHC social worker for case management. Standard care ranged from brief intervention by the SBHC social worker, to more intensive intervention by the SBHC social worker, to outside referral to local community service providers. SBHC social workers determined type and duration of services based on individual participant needs.
  Arms: Standard Care Control

SUMMARY:
The purpose of this study is to examine the efficacy of a culturally-grounded, school-based suicide and aggression preventive intervention for African American adolescents (Adapted-Coping with Stress Course [A-CWS]). The A-CWS is a 15-session, cognitive-behavioral group intervention designed to develop and enhance African American youths' skills for coping with stress. Emphasis is given to the identification of stress unique to the day-to-day experiences of the youths and options for reducing stress that are culturally consistent. A total of four public high schools in a large Midwestern metropolitan area participated in this study that used a randomized-controlled design, with randomization occurring at the individual level. Participants were randomized either to the A-CWS intervention condition, or to a standard care control condition. This study had three hypotheses: (1) The intervention would raise adaptive coping, relative to the standard care control condition; (2) coping skills would explain the effects of the A-CWS intervention on problematic outcomes (i.e., suicidality, aggression); and (3) socio-ecological factors (i.e., neighborhood and family characteristics) would influence the effect of the A-CWS intervention on coping skills, and the effect of coping skills on problematic outcomes.

DETAILED DESCRIPTION:
Participants were recruited from four urban, public schools, serving predominantly low-income, African American adolescents. Recruitment occurred over two years, with two cohorts of ninth-grade students recruited. Participants who returned student assent and active parent/guardian permission were screened for imminent suicide risk. Those participants who were identified as at imminent risk for suicide were referred to mental health professionals at the school-based health center for risk assessment and appropriate services. Participants not at imminent risk completed a baseline assessment of coping, aggression, and suicidality, and were randomly assigned to either the A-CWS intervention or standard care control conditions. Randomization occurred at the individual level.

Participants assigned to the A-CWS intervention condition received the 15-week A-CWS intervention. The intervention was facilitated by master's-level practitioners and implemented at the participating school during a non-instructional period of the school day. Intervention groups consisted of 8 to 10 participants, and intervention sessions were held for 45 minutes, once per week. Participants assigned to the standard care control condition were assigned to work with the school-based health center (SBHC) to receive standard behavioral services as delivered by SBHC mental health professionals.

To assess outcomes of adaptive coping, suicidality, and interpersonal aggression, participants were assessed at multiple timepoints. After completing a brief screening assessment, all participants, regardless of condition, were assessed a total of four times: (1) at baseline, prior to randomization, (2) immediately following the conclusion of the A-CWS intervention, (3) 6 months after the conclusion of the intervention, and (4) 12 months after the conclusion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled ninth-grade student, their parent/guardian, or primary teacher at participating school

Exclusion Criteria:

* Imminent suicide risk

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Suicide Ideation | Baseline, post-test, 6-month follow-up, 12-month follow-up
  Suicide ideation was measured with the Center for Epidemiological Studies - Depression (CES-D) Appended Suicide Measure, a 4-item self-report inventory that assesses suicide ideation during the last week.
Change in Aggression | Baseline, post-test, 6-month follow-up, 12-month follow-up
  Aggression was measured with a reduced 12-item version of the Aggression-Problem Behavior Frequency Scale, a self-report inventory that assesses the frequency of aggression in the last 30 days. This instrument has two subscales: physical aggression and non-physical aggression. Aggression was also measured using the Buss-Perry Aggression Questionnaire Short Form, a 12-item self-report inventory of aggression with four subscales: physical aggression, verbal aggression, anger, and hostility. In addition, aggression was measured with student behavioral data from participating schools, including number of detentions, suspensions, and reasons for detentions/suspensions. This data was used to identify the number of aggressive episodes per student and provided a secondary, archival measure of aggression.
Change in Coping | Baseline, post-test, 6-month follow-up, 12-month follow-up
  Coping was measured with a reduced 36-item version of the Adolescent Coping Orientation for Problem Experiences Measure, a self-report inventory that assesses frequency of use for coping methods used in response to stress. Seven subscales were included to assess preferred coping styles targeted by the intervention: ventilating feelings, seeking diversions, developing self-reliance, developing social support, investing in close friends, engaging in demanding activity, and relaxing.

CONTACTS AND LOCATIONS:
Overall Officials: LaVome Robinson, Ph.D., Principal Investigator — DePaul University
Locations (1):
- DePaul University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Robinson WL, Whipple CR, Keenan K, Flack CE, Lemke S, Jason LA. Reducing suicidal ideation in African American adolescents: A randomized controlled clinical trial. J Consult Clin Psychol. 2024 Feb;92(2):61-74. doi: 10.1037/ccp0000849. Epub 2023 Sep 28. PMID 37768628